CLINICAL TRIAL: NCT00938808
Title: Long-term Intervention With Weight Loss in Patients With Concomitant Obesity and Knee Osteoarthritis. The LIGHT Study
Acronym: LIGH T
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henning Bliddal (Other)
Collaborators: Velux Fonden (Other); Oak Foundation (Other); The Danish Rheumatism Association (Other); Cambridge Weight Plan Limited (Industry)
Responsible Party: Sponsor-Investigator, Henning Bliddal, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-B-2009-029
Record Dates: First submitted 2009-07-13; First posted 2009-07-14 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis, Knee; Obesity
Keywords: Osteoarthritis; Obesity; Weight loss; Dietary instruction; Formula diet; Attention
MeSH Terms: conditions — Osteoarthritis, Knee; Obesity; Osteoarthritis; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- One per day, Formula diet (Active Comparator): The Cambridge Programme. Formula diet One-daily
  Interventions: Dietary Supplement: day formula diet
- Repeated formula diet (Experimental): Dietary instruction (low-energy diet) 3x5 weeks per year
  Interventions: Dietary Supplement: day formula diet

INTERVENTIONS:
Dietary Supplement: day formula diet — The Cambridge Programme. Formula diet

SUMMARY:
Obesity and osteoarthritis (OA) co-exist in an increasing part of the population.

The two diseases intertwine in several ways. The evolution in the population shows a tendency towards deterioration of both by increasing general age and weight. The two diseases share pathogenetic features and the development of one disease increases the risk of the other and may be the onset of a vicious circle.

There is a link between treatments of these two diseases as well. There is now solid (gold) evidence that by treating effectively the obesity of patients with co-occurring OA, the functional status is dramatically ameliorated; the short-term results are equal to that of a joint replacement. The long-term efficacy of a weight loss remains to be shown. OA is definitely one of many diseases in which obesity must be taken seriously into account when planning a correct treatment of patients. This trial is an extension of the former CAROT trial NCT00655941. The participants of this trial are recruited for a prolongation of the dietary intervention consisting of a group therapy with low-energy diet in a randomized, two group (each n = 75 patients) study of maintenance of weight loss by continuing with supplementary either 3 x 5 weeks dietary supplements only or once-daily supplement. The hypothesis is that maintenance of the already induced weight loss is most efficiently ensured by the once-daily program.

DETAILED DESCRIPTION:
Any patient with osteoarthritis (OA) of the knee was invited to participate in the preceding trial. Eligible for this study will be patients, who have completed the one-year phase 2 of the CAROT. Exclusion criteria are planned knee alloplasty of both knees.

ELIGIBILITY:
Inclusion Criteria:

Former participant in the CAROT study ( NCT00655941 )

-

Exclusion Criteria:

Bilateral knee alloplasty -

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2009-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Weight, number of patients operated with knee alloplasty | 1 year, 3 years

SECONDARY OUTCOMES:
MRI | 1 year, 3 years
Gait analysis | 1 year, 3 years
Ultrasound | 1 year, 3 years
Collagen markers | 1 year, 3 years
Metabolic syndrome | 1 year, 3 years
KOOS | 1 year, 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, Professor, Principal Investigator — The P
Locations (1):
- The Parker Institute, Frederiksberg Hospital, Frederiksberg, Frederiksberg, Denmark

REFERENCES:
- [Background] Christensen R, Bartels EM, Astrup A, Bliddal H. Effect of weight reduction in obese patients diagnosed with knee osteoarthritis: a systematic review and meta-analysis. Ann Rheum Dis. 2007 Apr;66(4):433-9. doi: 10.1136/ard.2006.065904. Epub 2007 Jan 4. PMID 17204567
- [Background] Bliddal H, Christensen R. The management of osteoarthritis in the obese patient: practical considerations and guidelines for therapy. Obes Rev. 2006 Nov;7(4):323-31. doi: 10.1111/j.1467-789X.2006.00252.x. PMID 17038126
- [Background] Christensen R, Astrup A, Bliddal H. Weight loss: the treatment of choice for knee osteoarthritis? A randomized trial. Osteoarthritis Cartilage. 2005 Jan;13(1):20-7. doi: 10.1016/j.joca.2004.10.008. PMID 15639633
- [Derived] Christensen P, Henriksen M, Bartels EM, Leeds AR, Meinert Larsen T, Gudbergsen H, Riecke BF, Astrup A, Heitmann BL, Boesen M, Christensen R, Bliddal H. Long-term weight-loss maintenance in obese patients with knee osteoarthritis: a randomized trial. Am J Clin Nutr. 2017 Sep;106(3):755-763. doi: 10.3945/ajcn.117.158543. Epub 2017 Jul 26. PMID 28747328
- See also: Web page of the Parker Institute, Frederiksberg Hospital, Denmark — http://www.parkerinst.dk